CLINICAL TRIAL: NCT03987607
Title: Comparison of Electromyography-based TetraGraph and Acceleromyography-based TOF-Watch SX Neuromuscular Monitors Under Clinical Conditions
Brief Title: Comparison of Two Monitors That Measure Neuromuscular Function During Surgeries
Status: Completed | Type: Observational
Sponsor: Tamas Vegh, MD (Other)
Collaborators: Senzime AB (Industry)
Responsible Party: Sponsor-Investigator, Tamas Vegh, MD, associate professor, University of Debrecen
Organization: University of Debrecen (Other)
Other Study IDs: AITT2017/3
Record Dates: First submitted 2019-06-12; First posted 2019-06-17 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Neuromuscular Blockade
Keywords: neuromuscular monitoring; acceleromyography; electromyography
MeSH Terms: interventions — Neuromuscular Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patients scheduled for elective surgery: Patients scheduled for elective surgery requiring neuromuscular blockade
  Interventions: Device: neuromuscular blockade monitoring

INTERVENTIONS:
Device: neuromuscular blockade monitoring — Neuromuscular blockade monitoring via two different types of monitoring devices

SUMMARY:
Anesthesiologists are often required to give certain drugs, called muscle relaxants to the patients for surgery. These drugs make the people weak for the procedure to make the work of the surgeon easier and prevent unexpected movements. The effect of these drugs must be terminated by the end of the procedures to ensure that the patients can breathe normally. Over the years several monitors have been developed to monitor the effect of these drugs. The monitors use different principles to measure muscle function. Some monitors are integrated into anesthesia machines while others are battery-operated, portable devices. The aim of the present study is two compare monitors using different technologies. Both monitors stimulate a peripheral nerve at the wrist that makes the thumb twitch. The older device (TOF-Watch SX) measures the acceleration of thumb movement, the new device (TetraGraph) measures the electrical activity of the muscle that moves the thumb. The two devices will be connected so that with one simulation both types of signals can be recorded and analyzed. The monitors will be used during the surgeries as described by the manufacturer. The study will not influence the surgical procedure or the anesthetic of the patients. The aim of the study is to collect data on how the two monitors correlate, since they measure neuromuscular function by different technologies (acceleromyography and electromyography).

DETAILED DESCRIPTION:
The aim of this single center, one-arm, observational, prospective, non-inferiority study is to compare neuromuscular data obtained with two neuromuscular monitors. The two monitors are the electromyography-based TetraGraph neuromuscular monitor and the acceleromyography-based TOF-WATCH SX device.

The study will enroll 50 patients undergoing elective surgeries that require muscle relaxation. Patients will be only enrolled after written informed consent is obtained. Exclusion criteria include: neuromuscular disease in patient history, patient taking any medication that affects neuromuscular transmission, open wound or sores at the site of electrode placement, expected difficult airway, pregnancy or breastfeeding state, or implanted pacemaker.

The study will be conducted using one of the patient's arms. Both neuromuscular monitors will be applied on the same arm. The monitors will be connected by optical cable link to synchronize nerve stimulation and data recording. The aim of this setting is to obtain both acceleromyography and electromyography signals of the adductor pollicis muscle in response to ulnar nerve stimulation. This setting ensures identical stimulation conditions for the two monitors. Only the TOF-Watch SX will be used for nerve stimulation while the TOF-Watch will collect acceleromyography data of the thumb and TetraGraph will collect the electromyography data of the adductor pollicis muscle.

The ulnar nerve will be stimulated via single use electrocardiography electrodes used by TOF-Watch SX. The piezoelectric probe of TOF-Watch SX will be applied on the thumb via hand adapter, according to the manufacturer's instructions. The stimulating electrodes of TetraGraph will be isolated, since the device will not deliver electrical stimulation, only register the compound muscle action potentials of the adductor pollicis muscle evoked by TOF-Watch SX stimulation. The sensing electrodes of TetraGraph will be applied above the thenar and the interphalangeal joint of the thumb.

The TetraGraph monitor used for the study has a modified software compared to the commercially available monitors. This study device is used only for the current study.

Also, the cable of the TOF-Watch SX monitor has been modified to connect to the TetraGraph monitor for synchronization . The results of the responses analyzed by the TetraGraph device will not be used for clinical care decisions.

Neuromuscular monitoring will be started after the induction of anesthesia before the administration of neuromuscular blocking agent and terminated at the extubation of the patient. After calibration, the TOF-Watch will be left to stimulate automatically every 15 sec. Neuromuscular monitoring will be performed during surgery according to clinical standards, it will be stopped before extubation to avoid patient discomfort associated with neurostimulation.

During deep neuromuscular block the examiner will deliver post tetanic count stimulation every 5 min.

TOF-Watch SX data will be stored on a laptop computer using the devices software. TetraGraph is using a built-in SD card for data collection.

Beside acceleromyography and electromyography train-of-four ratios, train-of-four counts and post tetanic counts the following data will be recorded in a clinical research form:

* date of surgery, type of surgery,
* patient identification number, patient's sex, weight, height, BMI, dominant hand side,
* time of anesthesia induction, drugs used to induce anesthesia
* time of starting neuromuscular monitoring
* time of muscle relaxant administration, type and dose of muscle relaxant
* time of tracheal intubation and extubation,
* time of beginning and end of surgery
* time of reversal agent administration, type and dose of reversal agent
* use of surgical devices

To avoid uncertainty, only the data of TOF-Watch SX will be provided to the anesthesiology team for clinical use. TetraGraph data will be kept blinded from healthcare providers. All clinical decisions will be made according to TOF-Watch SX measurements, as per current clinical care. If any doubt arises regarding the reliability of the data delivered by TOF-Watch SX, the anesthesia workstations' built-in NMT modules (Infinity Trident NMT Smartpod, Draeger, Lübeck, Germany) will be used to guide clinical care.

Propofol target control infusion with bispectral index monitoring will be used to provide anesthesia. The administration of muscle relaxants, reversal agents and time of intubation and extubation will be at the discretion of the attending anesthesiologist as per usual clinical routine.

All patients will be monitored postoperatively for one day to detect any unexpected adverse events.

Statistical analysis:

Data will be analyzed offline after the completion of the study. Based on a priori sample size calculation, 50 patients will be enrolled in the study. Paired T-test and Bland-Altman analysis will be performed to examine the agreement between the two devices.

ELIGIBILITY:
Inclusion Criteria:

* elective surgery requiring neuromuscular blockade
* written informed consent
* American Society of Anesthesiology physical status I-III

Exclusion Criteria:

* neuromuscular disease in patient history,
* patient taking any medication that affects neuromuscular transmission,
* open wound or sores at the site of electrode placement,
* expected difficult airway,
* pregnancy or breastfeeding state,
* implanted pacemaker

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of the University of Debrecen Clinical Center who are scheduled for elective surgery
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2019-12-18 (Actual); Study Completion 2019-12-18 (Actual)

PRIMARY OUTCOMES:
Agreement between acceleromyography and electromyography derived TOF ratios in the recovery range of 0.8-1.0 | Prior to extubation
  Agreement between acceleromyography and electromyography derived TOF ratios in the recovery range of 0.8-1.0

SECONDARY OUTCOMES:
o Agreement between acceleromyography and electromyography derived TOF ratios in the recovery range of 0.6-0.79 | During surgery
  o Agreement between acceleromyography and electromyography derived TOF ratios in the recovery range of 0.6-0.79
o Agreement between acceleromyography and electromyography derived TOF ratios in the recovery range of 0.4-0.59 | During surgery
  o Agreement between acceleromyography and electromyography derived TOF ratios in the recovery range of 0.4-0.59
o Agreement between acceleromyography and electromyography derived TOF ratios in the recovery range of 0.2-0.39 | During surgery
  o Agreement between acceleromyography and electromyography derived TOF ratios in the recovery range of 0.2-0.39
o Agreement between acceleromyography and electromyography derived TOF counts | During surgery
  o Agreement between acceleromyography and electromyography derived TOF counts
o Agreement between acceleromyography and electromyography derived PTC counts | During surgery
  o Agreement between acceleromyography and electromyography derived PTC counts

CONTACTS AND LOCATIONS:
Locations (1):
- University of Debrecen, Department of Anesthesiology and Intensive Care, Debrecen, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liang SS, Stewart PA, Phillips S. An ipsilateral comparison of acceleromyography and electromyography during recovery from nondepolarizing neuromuscular block under general anesthesia in humans. Anesth Analg. 2013 Aug;117(2):373-9. doi: 10.1213/ANE.0b013e3182937fc4. Epub 2013 Jul 2. PMID 23821356
- [Background] Kopman AF, Chin W, Cyriac J. Acceleromyography vs. electromyography: an ipsilateral comparison of the indirectly evoked neuromuscular response to train-of-four stimulation. Acta Anaesthesiol Scand. 2005 Mar;49(3):316-22. doi: 10.1111/j.1399-6576.2005.00643.x. PMID 15752395
- [Background] Naguib M, Brull SJ, Johnson KB. Conceptual and technical insights into the basis of neuromuscular monitoring. Anaesthesia. 2017 Jan;72 Suppl 1:16-37. doi: 10.1111/anae.13738. PMID 28044330